CLINICAL TRIAL: NCT02469090
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Examine the Efficacy, Safety and Tolerability of APL-130277 in Levodopa Responsive Patients With Parkinson's Disease Complicated by Motor Fluctuations ("OFF" Episodes)
Brief Title: Efficacy, Safety and Tolerability Study of APL-130277 for the Acute Treatment of OFF Episodes in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTH-300
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Parkinson Disease, Off Episodes
Keywords: Parkinson Disease, off episodes
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APL-130277 (Experimental): APL-130277 sublingual thin film (10 mg, 15 mg, 20 mg, 25 mg, 30 mg and 35 mg)
  Interventions: Drug: APL-130277
- Placebo (Placebo Comparator): Matching placebo for APL-130277 sublingual thin film (10 mg, 15 mg, 20 mg, 25 mg, 30 mg and 35 mg)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APL-130277 — Use to treat up to 5 "OFF" episodes per day
  Other Names: Apomorphine Hydrochloride, Sublingual Thin Film
  Arms: APL-130277
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
A 12-week, prospective, multi-center, randomized, double-blind, placebo controlled, Phase 3 study in L-Dopa responsive PD patients with motor fluctuations ("OFF" episodes), designed to determine the efficacy, safety and tolerability of APL-130277.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Clinical diagnosis of Idiopathic PD, consistent with UK Brain Bank Criteria.
* Clinically meaningful response to L-Dopa with well-defined early morning "OFF" episodes, as determined by the Investigator.
* Receiving stable doses of L-Dopa/carbidopa (immediate or CR) administered at least 4 times per day OR Rytary™ administered 3 times per day, for at least 4 weeks before the initial Screening Visit
* No planned medication change(s) or surgical intervention anticipated during the course of study.
* Patients must experience at least one well defined "OFF" episode per day with a total daily "OFF" time duration of ≥ 2 hours during the waking day, based on patient self-assessment.
* Stage III or less on the modified Hoehn and Yahr scale in the "ON" state.
* MMSE score > 25.

Exclusion Criteria:

A patient will not be eligible for study entry if any of the following exclusion criteria are met:

* Atypical or secondary parkinsonism.
* Previous treatment with any of the following: a neurosurgical procedure for PD; continuous s.c. apomorphine infusion; or Duodopa/Duopa.
* Treatment with any form of s.c. apomorphine within 7 days prior to the initial Screening Visit (SV1). Patients that stopped s.c. apomorphine for any reason other than systemic safety concerns or lack of efficacy may be considered.
* Contraindications to APOKYN®, or hypersensitivity to apomorphine hydrochloride or any of the ingredients of APOKYN® (notably sodium metabisulfite); Tigan® (trimethobenzamide hydrochloride; patients from US sites only); or domperidone (patients from non-US sites only).
* Participation in a clinical trial within 30 days prior to the initial Screening Visit (SV1).
* Currently taking selective 5HT3 antagonists (i.e., ondansetron, granisetron, dolasetron, palonosetron, alosetron), dopamine antagonists (excluding quetiapine or clozapine) or dopamine depleting agents.
* Drug or alcohol dependency in the past 12 months.
* History of malignant melanoma.
* Clinically significant medical, surgical, or laboratory abnormality in the opinion of the Investigator.
* Major psychiatric disorder including, but not limited to, dementia, bipolar disorder, psychosis, or any disorder that, in the opinion of the Investigator, requires ongoing treatment that would make study participation unsafe or make treatment compliance difficult.
* History of clinically significant hallucinations during the past 6 months.
* History of clinically significant impulse control disorder(s).
* Dementia that precludes providing informed consent or would interfere with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (33):
- United States (32):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Muhammed Ali Parkinson and Movement Disorder CenterBarrow Neurological, Phoenix, Arizona
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - UC Irvine Health Gottschalk Medical Plaza, Irvine, California
  - Keck Medical Center at USC, Los Angeles, California
  - The Research Center of Southern California, Oceanside, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Parkinsons Disease and Movement Disorders Center, Boca Raton, Florida
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - USF Parkinson's Disease and Movement Disorder Center, Tampa, Florida
  - Emory University Department of Neurology, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Central DuPage Hospital - Neurodegenerative Clinic - Movement Disorders Center, Winfield, Illinois
  - Kansas University Medical Center - Department of Neurology, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - QUEST Research Institute, Farmington Hills, Michigan
  - Northern Michigan Neurology, Traverse City, Michigan
  - Henry Ford Hospital, West Bloomfield, Michigan
  - Columbia University Medical Center - Neurological Institute, Movement Disorders, New York, New York
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Jefferson University Hospital Philadelphia, Philadelphia, Pennsylvania
  - University of Virginia, Adult Neurology, Charlottesville, Virginia
  - Evergreen Health, Kirkland, Washington
- UHN Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Olanow CW, Factor SA, Espay AJ, Hauser RA, Shill HA, Isaacson S, Pahwa R, Leinonen M, Bhargava P, Sciarappa K, Navia B, Blum D; CTH-300 Study investigators. Apomorphine sublingual film for off episodes in Parkinson's disease: a randomised, double-blind, placebo-controlled phase 3 study. Lancet Neurol. 2020 Feb;19(2):135-144. doi: 10.1016/S1474-4422(19)30396-5. Epub 2019 Dec 7. PMID 31818699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with Levodopa (L-dopa) responsive idiopathic Parkinson's Disease (PD) complicated by motor fluctuations ('OFF' episodes) were recruited in 33 study sites in the United States and Canada starting June 2015. Study completed in December 2017. Approval was obtained from the Enrollment Adjudication Committee prior to enrollment of each patient.
Pre-assignment Details: The study included a Dose Titration Phase in which individual responses to single doses of APL-130277 (10 - 35 milligram [mg]) were evaluated at 5 mg dose increments to determine the starting dose that achieved a full 'ON' within 45 minutes. Patients were randomized at this dose to APL-130277 or placebo in the 12-week Maintenance Treatment Phase.
Groups:
- APL-130277 (Titration): Patients were titrated to identify the efficacious and tolerable dose of APL-130277.
  On Titration Visit 1 (TV1), patients presented to the clinic in an 'OFF' state and received 10 mg APL-130277. Patients who responded to 10 mg APL-130277 with a full 'ON' response within 45 minutes of dosing, as assessed by the patient and Investigator, completed the Dose Titration Phase.
  If a complete 'ON' response was not achieved within 45 minutes of dosing, patients restarted their normal PD medication and returned to the clinic within 3 days for the next TV, to receive the next sequential dose of APL-130277 (15 mg at TV2, 20 mg at TV3, 25 mg at TV4, 30 mg at TV5 and 35 mg at TV6). Patients who achieved a full 'ON' response within 45 minutes at a given dose were randomized to the Maintenance Treatment Phase. Any patients who reached 35 mg at TV6 and did not exhibit a full 'ON' response were discontinued.
- Placebo (Maintnance): Patients who completed the Dose Titration Phase and were randomized in a blinded manner (1:1 ratio) to receive placebo in the 12-week double-blind Maintenance Treatment Phase. Patients self-administered the matching placebo for the strength of treatment determined during the Dose Titration Phase in up to 5 'OFF' episodes per day for 12 weeks in the at-home portion of the study. Patients returned to the clinic in 4-week intervals for safety and efficacy assessments. Patients completed a dosing diary at home for 2 days prior to the scheduled visit.
- APL-130277 (Maintenance): Patients who completed the Dose Titration Phase and were randomized in a blinded manner (1:1 ratio) to receive APL-130277 in the 12-week double-blind Maintenance Treatment Phase. Patients self-administered the strength of treatment determined during the Dose Titration Phase in up to 5 'OFF' episodes per day for 12 weeks in the at-home portion of the study. Patients returned to the clinic in 4-week intervals for safety and efficacy assessments. Patients completed a dosing diary at home for 2 days prior to the scheduled visit.
Period: Period 1: Dose Titration Phase
Arm/Group | APL-130277 (Titration) | Placebo (Maintnance) | APL-130277 (Maintenance)
Started | 141 | 0 | 0
Completed | 109 | 0 | 0
Not Completed | 32 | 0 | 0
Not completed — Adverse Event | 12 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 11 | 0 | 0
Period: Period 2: Maintenance Treatment Phase
Arm/Group | APL-130277 (Titration) | Placebo (Maintnance) | APL-130277 (Maintenance)
Started | 0 (Subjects who completed the Titration Phase were eligible to proceed to Maintenance Treatment Phase) | 55 (subjects who completed the Titration Phase and were randomized to Placebo in the Maintenance Phase) | 54 (subjects who completed the Titration Phase and were randomized to APL-130277 Maintenance Phase)
Completed | 0 | 46 | 34
Not Completed | 0 | 9 | 20
Not completed — Adverse Event | 0 | 5 | 15
Not completed — Withdrawal by Subject | 0 | 3 | 4
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo (Maintenance): Patients who completed the Dose Titration Phase and were randomized in a blinded manner (1:1 ratio) to receive placebo in the 12-week double-blind Maintenance Treatment Phase. Patients self-administered the matching placebo for the strength of treatment determined during the Dose Titration Phase in up to 5 'OFF' episodes per day for 12 weeks in the at-home portion of the study. Patients returned to the clinic in 4-week intervals for safety and efficacy assessments. Patients completed a dosing diary at home for 2 days prior to the scheduled visit.
- APL-130277 (Mainenance): Patients who completed the Dose Titration Phase and were randomized in a blinded manner (1:1 ratio) to receive APL-130277 in the 12-week double-blind Maintenance Treatment Phase. Patients self-administered the strength of treatment determined during the Dose Titration Phase in up to 5 'OFF' episodes per day for 12 weeks in the at-home portion of the study. Patients returned to the clinic in 4-week intervals for safety and efficacy assessments. Patients completed a dosing diary at home for 2 days prior to the scheduled visit.
- Total: Total of all reporting groups
Arm/Group | Placebo (Maintenance) | APL-130277 (Mainenance) | Total
Number analyzed (Participants) | 55 | 54 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 30 | 64
  >=65 years | 21 | 24 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 17 | 41
  Male | 31 | 37 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 52 | 51 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 0 | 2
  White | 51 | 50 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 53 | 108
  Canada | 0 | 1 | 1
Time Since Diagnosis of PD [Mean (Standard Deviation); unit: years] | 9.3 (3.84) | 8.7 (4.25) | 9.0 (4.04)
Time Since Motor Fluctuations Started [Mean (Standard Deviation); unit: years] | 4.54 (3.780) | 4.69 (3.916) | 4.61 (3.831)
Type of 'OFF' episodes experienced [Number; unit: participants]
  Morning akinesia | 44 | 46 | 90
  Wearing "OFF" | 54 | 54 | 108
  Delayed "ON" | 43 | 29 | 72
  Dose Failure | 23 | 22 | 45
  Sudden :OFF" | 32 | 26 | 58
Number of 'OFF' Episodes Typically Experienced Per Day [Mean (Standard Deviation); unit: "OFF" episodes/day] | 3.8 (1.40) | 3.9 (1.17) | 3.9 (1.29)
Length of 'OFF' Episodes [Mean (Standard Deviation); unit: Minutes] | 66.1 (30.09) | 63.7 (31.91) | 64.9 (30.89)
ON' State Modified Hoehn and Yahr Score [Number; unit: participants] — The Modified Hoehn and Yahr Scale was used to assess the patient's motor function during screening.
  0 = Asymptomatic, 1 = Unilateral involvement only, 1.5 = Unilateral and axial involvement, 2 = Bilateral involvement without impairment of balance, 2.5 = Mild bilateral disease with recovery on pull test, 3 = Mild to moderate involvement; some postural instability but physically independent; needs assistance to recover from pull test, 4 = Severe disability; still able to walk or stand unassisted, 5 = Wheelchair bound or bedridden unless aided.
  participants
    Hoehn and Yahr Score = 0 | 0 | 0 | 0
    Hoehn and Yahr Score = 1 | 1 | 0 | 1
    Hoehn and Yahr Score = 1.5 | 0 | 0 | 0
    Hoehn and Yahr Score = 2 | 38 | 41 | 79
    Hoehn and Yahr Score = 2.5 | 4 | 8 | 12
    Hoehn and Yahr Score = 3 | 11 | 5 | 16
    Hoehn and Yahr Score = 4 | 0 | 0 | 0
    Hoehn and Yahr Score = 5 | 0 | 0 | 0
    Missing | 1 | 0 | 1
Total Daily L-Dopa Dose [Mean (Standard Deviation); unit: mg] | 1007.73 (562.323) | 1058.70 (563.301) | 1032.98 (560.781)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Pre-Dose to 30 Minutes Post-Dose in The Movement Disorders Society Unified Parkinson's Disease Rating Scale Part III Motor Examination (MDS-UPDRS Part III) Score at Maintenance Visit 4 (MV4) - Week 12
Description: The Motor Function section (Part III) of the MDS-UPDRS was administered by the Investigator, and included 33 scores based on 18-items, each anchored with 5 responses: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range was from 0 to 132, with a lower score indicating better motor function and a higher score indicating more severe motor symptoms.
  The least square mean change in the MDS-UPDRS Part III score from pre-dose to 30 minutes post-dose at MV4 is presented. A negative change from pre-dose indicates an improvement.
Time Frame: At t=0 (just prior to dosing) and t=30 minutes at MV4 (Week 12 of the Maintenance Treatment Phase).
Population: The modified Intention-To-Treat (mITT) Population consisted of all patients who were randomized and received at least 1 post-randomization dose of study medication (APL-130277 or placebo). Patients were grouped according to the randomized treatment group. Only patients with data available for analysis at the time point are presented.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 55 | 54
Units on a scale | -3.5 (1.29) | -11.1 (1.46)
Statistical Analysis 1: Comparison: Placebo (Maintenance) vs APL-130277 (Maintenance); Mixed effects model for repeated measures (MMRM) was used to estimate the treatment difference(APL-130277-placebo) Observed change from pre-dose MDS-UPDRS Part III score values after 30 minutes were response values. Treatment group, visit and the interaction between the treatment group and visit were fixed factors. Change from pre-dose in MDS-UPDRS Part III score after 30 minutes at the last TV at which the randomized dose was given up through TV6 was used as a covariate; Test type: Superiority; p = 0.0002, LS mean difference — The null-hypothesis to be tested was: H0: APL-130277 is the same as placebo in its effect on the motor function against the 2-sided alternative: H1: Either of the treatment groups is superior to the other in its effect on the motor function; To control the family-wise type I error rate, the primary and secondary end points were tested in hierarchical order in the order presented; LS mean differnce = -7.6, 95% CI 2-sided [-11.5 to -3.7], Standard Error of Mean 1.96

2. Secondary Outcome: Percentage of Patients With a Patient-related Full 'ON' Response Within 30 Minutes at MV4 - Week 12: Predicted Response Rate
Description: A full 'ON' response was defined as a period of time where in the judgment of the patient the medication was providing full benefit with regard to mobility, stiffness, slowness and other PD features comparable to or better than that obtained with their standard dose of oral L-dopa and other anti-parkinsonian medications prior to beginning the study. Patients were asked if they attained a full 'ON' state anytime within 30 minutes of dosing. The predicted response rates are presented and were estimated using a generalized linear mixed model.
Time Frame: At t=30 minutes at MV4 (Week 12 of the Maintenance Treatment Phase).
Population: The mITT Population consisted of all patients who were randomized and received at least 1 post-randomization dose of study medication (APL-130277 or placebo). Patients were grouped according to the randomized treatment group. Only patients with data available for analysis at the time point are presented.
Measure: Number; unit: number of participants
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 55 | 54
number of participants | 16 | 35
Statistical Analysis 1: Comparison: Placebo (Maintenance) vs APL-130277 (Maintenance); This was analyzed using a generalized linear mixed model (with logit link function) for binomial data. The model included the observed outcomes as the response values, with treatment group, visit, and the interaction between treatment group and visit as fixed factors and the "ON/OFF" assessment at the last open-label titration visit at which the randomized dose was given as a covariate; Test type: Superiority; p = 0.0426, Adjusted Odds Ratio; Adjusted odds ratio = 2.81, 95% CI 2-sided [1.036 to 7.644]

3. Secondary Outcome: Percentage of Patients With a Patient-related Full 'ON' Response Within 30 Minutes That Had a Duration of Effect of at Least 30 Minutes at MV4 - Week 12: Predicted Response Rate
Description: A full 'ON' response was defined as a period of time where in the judgment of the patient the medication was providing full benefit with regard to mobility, stiffness, slowness and other PD features comparable to or better than that obtained with their standard dose of oral L-dopa and other anti-parkinsonian medications prior to beginning the study. The percentage of patients who attained a full 'ON' within 30 minutes of dosing, and whose duration from time when study medication began to have an effect lasted for at least 30 minutes were evaluated. The predicted response rates are presented and were estimated using a generalized linear mixed model.
Time Frame: At MV4 (Week 12 of the Maintenance Treatment Phase).
Population: as for outcome 2
Measure: Number; unit: number of participants
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 55 | 54
number of participants | 14 | 31
Statistical Analysis 1: Comparison: Placebo (Maintenance) vs APL-130277 (Maintenance); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0501, Adjusted odds ratio — The hierarchical testing stopped at this endpoint due to non-significant result. P-values for endpoints after this endpoint have not been presented and the confidence interval presented are unadjusted for multiplicity; Adjusted odds ratio = 2.80, 95% CI 2-sided [1.00 to 7.84]

4. Secondary Outcome: Patient Global Impression of Improvement (PGI-I): Percentage of Patients Who Improved at MV4 - Week 12
Description: During the PGI-I assessment the patient was asked to answer the question "Since starting study medication, how has your illness changed?" with 1 of the following responses:
  1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse and 7 = very much worse.
  The percentage of patients who improved at MV4 (gave responses 1 - 3) are presented.
Time Frame: At MV4 (Week 12 of the Maintenance Treatment Phase).
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 55 | 54
percentage of participants | 20.0 | 37.0

5. Secondary Outcome: Clinician Global Impression of Improvement (CGI-I): Percentage of Patients Who Improved at MV4 - Week 12
Description: During the CGI-I assessment the clinician using the question "Compared to his/her condition on baseline, how much has he/she changed?" provided 1 of the following responses:
  1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse and 7 = very much worse.
  The percentage of patients who improved at MV4 (responses 1 - 3) are presented.
Time Frame: At MV4 (Week 12 of the Maintenance Treatment Phase).
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 55 | 54
percentage of participants | 20.0 | 40.7

6. Secondary Outcome: Mean Change From Screening Visit to MV4 (Week 12) in MDS-UPDRS Part II: Motor Aspects of Experience of Daily Living
Description: Part II of the MDS-UPDRS assessed motor experiences of daily living and was self-administered by the patient. The MDS-UPDRS Part II score was calculated as the sum of the individual items of the MDS-UPDRS Part II questionnaire (items 2.1 - 2.13), and was based on 13-items, each anchored with 5 responses: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range was from 0 to 52, with a lower score indicating better motor function for daily living and a higher score indicating more severe motor symptoms.
  The mean change in the MDS-UPDRS Part II score from the screening visit to Week 12 of the Maintenance Treatment Phase is presented. A negative change indicates an improvement.
Time Frame: At Screening Visit and at MV4 (Week 12 of the Maintenance Treatment Phase).
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 44 | 33
units on a scale | 2.095 [0.749 to 3.440] | 0.995 [-0.559 to 2.549]
Statistical Analysis 1: Comparison: Placebo (Maintenance) vs APL-130277 (Maintenance); Test type: Superiority; LS mean difference = -1.100, 95% CI 2-sided [-3.159 to 0.959]

7. Secondary Outcome: Mean Percentage of Instances Where a Full 'ON' Response Was Achieved at 30 Minutes Post-dose on the Home Dosing Diary Entries During the 2 Days Prior to MV4 - Week 12
Description: Patients self-administered their doses of randomized study medication in order to treat up to 5 'OFF' episodes per day and recorded the time of self-administration and the 'ON'/'OFF' status at 30 minutes post-dose in a home dosing diary.
  A full 'ON' response was defined as a period of time where in the judgment of the patient the medication was providing full benefit with regard to mobility, stiffness, slowness and other PD features comparable to or better than that obtained with their standard dose of oral L-dopa and other anti-parkinsonian medications prior to beginning the study.
  The percentage of instances in which a full 'ON' response was achieved at 30 minutes out of all recorded episodes was calculated and is presented, and the mean percentage is presented.
Time Frame: 2 days prior to MV4 (Week 12 of the Maintenance Treatment Phase).
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of instnces
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 55 | 54
percentage of instnces | 31.10 [19.25 to 42.95] | 78.70 [64.16 to 93.24]
Statistical Analysis 1: Comparison: Placebo (Maintenance) vs APL-130277 (Maintenance); Test type: Superiority; LS mean difference = 47.60, 95% CI 2-sided [28.84 to 66.36]

8. Secondary Outcome: Mean Change From Screening Visit to MV4 in the Parkinson's Disease Quality of Life Questionnaire (PDQ-39) Summary Index Score
Description: The PDQ-39 was self-administered by the patient during screening and at each MV. The PDQ-39 assessed the impact of PD on the quality of life in the preceding month using 39-items, each anchored with 5 responses: Never, Occasionally, Sometimes, Often and Always. Items were grouped into 8 scales (Mobility, Activities of daily living, Emotional well-being, Stigma, Social support, Cognitions, Communication and Bodily discomfort) that were scored by expressing summed item scores as a percentage score ranging between 0 and 100. The PDQ-39 summary index score was derived by the sum of the 8 PDQ-39 scale scores divided by 8, yielding a score between 0 and 100. 0 indicates perfect health and 100 indicates worse health as assessed by the measure. A negative change indicates an improvement.
Time Frame: At Screening Visit and at MV4 (Week 12 of the Maintenance Treatment Phase).
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 55 | 54
units on a scale | -1.671 [-4.442 to 1.101] | 0.309 [-2.748 to 3.366]
Statistical Analysis 1: Comparison: Placebo (Maintenance) vs APL-130277 (Maintenance); Test type: Superiority; LS mean difference = 1.979, 95% CI 2-sided [-2.162 to 6.120]

9. Secondary Outcome: Mean Change From Pre-Dose to 15 Minutes Post-Dose in the MDS-UPDRS Part III Score at MV4 - Week 12
Description: The Motor Function section (Part III) of the MDS-UPDRS was administered by the Investigator, and included 33 scores based on 18-items, each anchored with 5 responses: 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range was from 0 to 132, with a lower score indicating better motor function and a higher score indicating more severe motor symptoms.
  The mean change in the MDS-UPDRS Part III score from pre-dose to 15 minutes post-dose at MV4 is presented. A negative change indicates an improvement.
Time Frame: At t=0 (just prior to dosing) and t=15 minutes at MV4 (Week 12 of the Maintenance Treatment Phase).
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 55 | 54
units on a scale | -3.0 [-5.1 to -0.8] | -6.4 [-8.8 to -4.0]
Statistical Analysis 1: Comparison: Placebo (Maintenance) vs APL-130277 (Maintenance); Test type: Superiority; LS mean difference = -3.4, 95% CI 2-sided [-6.7 to -0.2]

10. Secondary Outcome: Time From Dosing to When Study Medication Provided an Effect at MV4 - Week 12
Description: The time to effect at MV4 was described using the Kaplan-Meier method, including an estimate of the median time to effect and corresponding 95% confidence interval.
Time Frame: At MV4 (Week 12 of the Maintenance Treatment Phase).
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo (Maintenance) | APL-130277 (Maintenance)
Number analyzed (Participants) | 55 | 54
Minutes | NA [42.73 to NA] — Less than 40% of placebo patients were observed to have the event. | 21.2 [15.00 to 27.00]
Statistical Analysis 1: Comparison: Placebo (Maintenance) vs APL-130277 (Maintenance); Median Time to effect for APL-130277 versus placebo patients; Test type: Superiority; Hazard ratio = 3.4, 95% CI 2-sided [1.99 to 5.69]

ADVERSE EVENTS:
Time Frame: Dose Titration Phase (21 days): all AEs that started on/after the first dose of APL-130277 but before the first dose of study medication during the Maintenance Treatment Phase. Maintenance Treatment Phase (12 weeks): all AEs that started on/after the first dose of study medication during the Maintenance Treatment Phase.
Description: All AEs were collected for each patient. Patients were queried in a non-leading manner, without specific prompting. Treatment emergent AEs are presented for the Dose Titration Phase (APl-130277 [titration]) and for the Maintenance Treatment Phase (APL-130277 [maintenance] and Placebo [maintenance]).
Arm/Group | APL-130277 (Titration) | Placebo (Maintenance) | APL-130277 (Maintenance)
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/55 | 1/54
Serious Adverse Events (participants affected / at risk) | 1/141 | 1/55 | 2/54
Other Adverse Events (participants affected / at risk) | 60/141 | 12/55 | 39/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APL-130277 (Titration) (N=141) | Placebo (Maintenance) (N=55) | APL-130277 (Maintenance) (N=54)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than .03% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APL-130277 (Titration) (N=141) | Placebo (Maintenance) (N=55) | APL-130277 (Maintenance) (N=54)
Nausea (Gastrointestinal disorders) | 29 (40) | 2 (2) | 15 (18)
Oral mucosalerythema (Gastrointestinal disorders) | 6 (13) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 6 (6) | 0 (0) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 2 (4) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Lip oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Lip ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 16 (28) | 1 (1) | 7 (11)
Dizziness (Nervous system disorders) | 16 (21) | 0 (0) | 5 (6)
Headache (Nervous system disorders) | 11 (16) | 0 (0) | 3 (3)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Yawning (Respiratory, thoracic and mediastinal disorders) | 17 (27) | 1 (1) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (16) | 0 (0) | 4 (5)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Chills (General disorders) | 8 (11) | 0 (0) | 2 (3)
Fatigue (General disorders) | 4 (4) | 0 (0) | 4 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (9) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (4)
Anxiety (Psychiatric disorders) | 4 (5) | 1 (1) | 2 (2)
Flushing (Vascular disorders) | 4 (7) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites,Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT02469090/SAP_000.pdf
  • Study Protocol (2015-05-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT02469090/Prot_001.pdf